CLINICAL TRIAL: NCT00927472
Title: A Multi-Center Phase III Study to Evaluate Ovide Lotion 0.5% Formulation, for the Control of Head Lice in Pediatric Subjects and Adult Subjects With Pediculosis Capitis
Brief Title: Efficacy, Safety and Tolerability of a Novel Malathion Formulation in Patients 2 Years and Older With Head Lice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MALG-0817
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Pediculosis
Keywords: Head Lice
MeSH Terms: conditions — Lice Infestations | interventions — Permethrin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Malathion Gel (Experimental): Malathion gel 0.5% 30 minute application
  Interventions: Drug: Malathion gel 0.5%
- Nix Creme Rinse (Active Comparator): Nix applied to scalp for 10 minutes
  Interventions: Drug: Permethrin 1% rinse

INTERVENTIONS:
Drug: Malathion gel 0.5% — Malathion gel 0.5% applied to scalp for 30 minutes. May be repeated in 1 week if head lice are still present.
  Arms: Malathion Gel
Drug: Permethrin 1% rinse — Permethrin 1% shampooed into scalp for 10 minutes. May be repeated in 1 week if head lice are still present.
  Other Names: Nix Creme Rinse
  Arms: Nix Creme Rinse

SUMMARY:
In this study, Malathion Gel 0.5% will be compared to Nix (permethrin 1%) as a treatment for head lice in patients 2 years of age and older. Malathion Gel 0.5% is a new formulation of an established head lice treatment. The new formulation has been evaluated in 2 previous studies of patients 2 years of age and older.

DETAILED DESCRIPTION:
This is a Phase III, multi-center, investigator-blinded, two-arm, randomized, parallel group study, evaluating the safety and efficacy of a Malathion Gel, 0.5% formulation, manufactured by Taro. The objective is to show superiority of the novel product to an active control, Nix® Crème Rinse, manufactured by Insight Pharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed active head lice infestation

Exclusion Criteria:

* Allergy to pediculicides or hair care products
* Scalp conditions other than head lice
* Previous head lice treatment within the past 4 weeks
* Current antibiotic treatment

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Investigator Site, Bentonville, Arkansas
  - Investigator Site, Jonesboro, Arkansas

REFERENCES:
- [Background] Meinking TL, Vicaria M, Eyerdam DH, Villar ME, Reyna S, Suarez G. A randomized, investigator-blinded, time-ranging study of the comparative efficacy of 0.5% malathion gel versus Ovide Lotion (0.5% malathion) or Nix Creme Rinse (1% permethrin) used as labeled, for the treatment of head lice. Pediatr Dermatol. 2007 Jul-Aug;24(4):405-11. doi: 10.1111/j.1525-1470.2007.00460.x. PMID 17845167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 2 dermatology clinical practices
Period: Overall Study
Arm/Group | Malathion Gel | Nix Creme Rinse
Started | 126 | 128
Completed | 115 | 106
Not Completed | 11 | 22
Not completed — Withdrawal by Subject | 10 | 11
Not completed — Lost to Follow-up | 1 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Post treatment Assessment out of window | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were evaluated to identify differences between treatment groups which were not eliminated by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Malathion Gel | Nix Creme Rinse | Total
Number analyzed (Participants) | 126 | 128 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.91 (11.79) | 14.02 (11.88) | 13.96 (11.68)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 95 | 97 | 192
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 104 | 205
  Male | 25 | 24 | 49
Region of Enrollment [Number; unit: participants]
  United States | 126 | 128 | 254

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Index Subjects Free of Any of Lice 14 Days After Their Last Treatment.
Description: Treatment Success was evaluated using the Efficacy Intention to Treat (eITT) (LOCF) Efficacy ITT (eITT) was considered definitive.
  The primary efficacy variable was the proportion of index subjects who were considered a Treatment Success 14 days after their last treatment (Day 14 visit if only treated on Day 1, Day 21 visit if treated on Day 1 and Day 7).
  Index subject: 95 from 254 randomized (the youngest subject in the household who met index case criteria( having nits and at least 3 live lice))
Time Frame: 3 weeks
Population: The Efficacy Intention to Treat (eITT) population was the primary population for demonstrating the superiority of the Malathion product to the active control Nix® Crème Rinse.
  eITT population: included all index subjects with at least one application of treatment.
  Proportion of Subjects that are lice-free 14 days after their last treatment
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 47 | 48
percentage of subjects | 82.98 (3.25) | 62.50 (4.95)
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.0386, t-test, 2 sided

2. Secondary Outcome: Proportion of Subjects Who Were Considered Treatment Success 14 Days After Their First Treatment in the Efficacy ITT (LOCF))
Description: Treatment Success in the Efficacy ITT (LOCF)
  The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
Time Frame: 3 weeks
Population: Treatment Success in the Efficacy ITT (LOCF). The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment. Based on the protocol predefined imputation of missing efficacy data, the effective sample size = 82; frequency missing = 13.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 42 | 40
percentage of subjects | 80.95 | 70.00
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.3675, t-test, 2 sided

3. Primary Outcome: Proportion of Index Subjects Lice-free 2 Weeks After Their Last Treatment
Description: Treatment Success in the Efficacy Intention to Treat (eITT) (No LOCF)
  The primary efficacy variable was the proportion of index subjects who were considered a Treatment Success 14 days after their last treatment (Day 14 visit if only treated on Day 1, Day 21 visit if treated on Day 1 and Day 7).
Time Frame: 3 weeks
Population: Treatment Success in the Efficacy ITT (No LOCF) The Efficacy ITT population was the primary population for demonstrating the superiority of the Malathion product to the active control Nix® Crème Rinse.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 47 | 48
percentage of subjects | 78.72 | 58.33
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.0490, t-test, 2 sided

4. Primary Outcome: Proportion of Index Subjects Lice-free 14 Days After Their Last Treatment
Description: Treatment Success in the Per Protocol Population (PPP)
  The PPP included all subjects who complied strictly with the protocol and had outcome data for all required visits. Superiority analysis in the PPP was considered to be supportive.
Time Frame: 3 weeks
Population: The Per-Protocol Population (PPP) included all subjects who complied strictly with the protocol and had outcome data for all required visits. Superiority analysis in the PPP was considered to be supportive.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 115 | 106
percentage of subjects | 91.30 | 71.70
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

5. Primary Outcome: Proportion of All Randomized Subjects Who Were Treated and Returned for at Least One Post-treatment Visit.(LOCF)
Description: Treatment Success in the Modified Intention to Treat (Modified ITT) (LOCF)
  The Modified ITT included all randomized subjects who were treated and returned for at least one post-treatment visit. Subjects with missing efficacy data were included first with LOCF and then with non-LOCF
Time Frame: 3 weeks
Population: Treatment Success in the Modified Intention to Treat ( Modified ITT) (LOCF) The Modified ITT included all randomized subjects who were treated and returned for at least one post-treatment visit. Subjects with missing efficacy data were included first with LOCF and then with non-LOCF.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 121 | 111
percentage of subjects | 91.74 | 72.97
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided

6. Primary Outcome: Proportion of All Randomized Subjects Who Were Treated and Returned for at Least One Post-treatment Visit (Non-LOCF).
Description: Treatment Success in the Modified ITT (non-LOCF)
  The Modified ITT included all randomized subjects who were treated and returned for at least one post-treatment visit.
  Subjects with missing efficacy data were included first with LOCF and then with non-LOCF
Time Frame: 3 weeks
Population: Treatment Success in the Modified ITT (LOCF) The Modified ITT included all randomized subjects who were treated and returned for at least one post-treatment visit. Subjects with missing efficacy data were included first with LOCF and then with non-LOCF.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 121 | 111
percentage of subjects | 86.78 | 68.47
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.0012, t-test, 2 sided

7. Secondary Outcome: Proportion of Subjects Who Were Considered Treatment Success 14 Days After Their First Treatment in the Efficacy ITT (Non LOCF))
Description: Treatment Success in the Efficacy ITT (non LOCF)
  The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
Time Frame: 3 weeks
Population: Treatment Success was evaluated in the Efficacy ITT(non LOCF) The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
  Based on the protocol predefined imputation of missing efficacy data, the effective sample size = 82; frequency missing = 13.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 42 | 40
percentage of subjects | 76.19 | 65.00
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.3817, t-test, 2 sided

8. Secondary Outcome: Proportion of Subjects Who Were Considered Treatment Success 14 Days After Their First Treatment in the PPP
Description: Treatment Success in the PPP
  The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
  The evaluations in the PPP was considered supportive.
Time Frame: 3 weeks
Population: The evaluations in the PPP was considered supportive The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
  Based on the protocol predefined imputation of missing efficacy data, the effective sample size = 188; frequency missing = 33.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 104 | 84
percentage of subjects | 90.38 | 80.95
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.1059, t-test, 2 sided

9. Secondary Outcome: Proportion of Subjects Who Were Considered Treatment Success 14 Days After Their First Treatment in the Modified ITT (LOCF)
Description: Treatment Success in the Modified ITT (LOCF)
  The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
  The evaluations in the Modified ITT was considered supportive.
Time Frame: 3 weeks
Population: The evaluations was in the Modified ITT was considered supportive. The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
  Based on the protocol predefined imputation of missing efficacy data, the effective sample size = 199; frequency missing = 33.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 110 | 89
percentage of subjects | 90.91 | 82.02
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.1088, t-test, 2 sided

10. Secondary Outcome: Proportion of Subjects Who Were Considered Treatment Success 14 Days After Their First Treatment in the Modified ITT (Non LOCF)
Description: Treatment Success in the Modified ITT (non LOCF)
  The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
  The evaluations in the Modified ITT was considered supportive.
Time Frame: 3 weeks
Population: The evaluations in the Modified ITT was considered supportive. The secondary efficacy variable was the proportion of index subjects who were lice-free 14 days after their first treatment.
  Based on the protocol predefined imputation of missing efficacy data, the effective sample size = 199; frequency missing = 33.
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Creme Rinse
Number analyzed (Participants) | 110 | 89
percentage of subjects | 85.45 | 76.40
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Creme Rinse; Test type: Superiority or Other; p = 0.1527, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Malathion Gel | Nix Creme Rinse
Serious Adverse Events (participants affected / at risk) | 1/126 | 0/128
Other Adverse Events (participants affected / at risk) | 20/126 | 8/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Malathion Gel (N=126) | Nix Creme Rinse (N=128)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.79% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Malathion Gel (N=126) | Nix Creme Rinse (N=128)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 3 (3) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 6 (7) | 0 (0)
Application site oedema (General disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2)
Chemical eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Scratch (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No